CLINICAL TRIAL: NCT07348198
Title: Histologic and Histomorphometric Evaluation of Lateral Maxillary Sinus Augmentation Using Demineralized Freeze-Dried Bone Allograft With or Without Platelet-Rich Fibrin: A Prospective Split-Mouth Clinical Study
Brief Title: Histologic and Histomorphometric Evaluation of Lateral Maxillary Sinus Augmentation With or Without Platelet-Rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Erkin Doğan, Research Assistant, Marmara University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Biruni Uni. 2015-KAEK-76-23-07
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Sinus Augmentation; Posterior Maxillary Atrophy
Keywords: sinus augmentation; Split-mouth design; Platelet-rich fibrin; Histomorphometric analysis; Dental implants; demineralized freeze-dried bone allograft
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, split-mouth (within-subject) clinical trial in which each participant receives both interventions on contralateral maxillary sinuses.
Who Masked: Outcomes Assessor
Masking Description: Histological and histomorphometric analyses were performed by a blinded examiner who was unaware of the intervention allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non- PRF(DFDBA Alone) (Experimental): Lateral maxillary sinus augmentation performed using demineralized freeze-dried bone allograft (DFDBA) alone.
  Interventions: Procedure: Lateral Maxillary Sinus Augmentation With DFDBA
- PRF(DFDBA + PRF) (Experimental): Lateral sinus floor elevation using demineralized freeze-dried bone allograft combined with autologous platelet-rich fibrin.
  Interventions: Procedure: Lateral Maxillary Sinus Augmentation With DFDBA and PRF

INTERVENTIONS:
Procedure: Lateral Maxillary Sinus Augmentation With DFDBA — Lateral sinus floor elevation using demineralized freeze-dried bone allograft for bone augmentation prior to implant placement.
  Arms: Non- PRF(DFDBA Alone)
Procedure: Lateral Maxillary Sinus Augmentation With DFDBA and PRF — Lateral sinus floor elevation using demineralized freeze-dried bone allograft combined with autologous platelet-rich fibrin.
  Arms: PRF(DFDBA + PRF)

SUMMARY:
This study evaluates bone healing after lateral maxillary sinus lift surgery performed prior to dental implant placement. This surgical procedure is commonly used when there is insufficient bone height in the upper jaw to support dental implants.

Patients who required sinus lift surgery on both sides of the upper jaw were included in the study. In each patient, one side was treated with a demineralized freeze-dried bone allograft (DFDBA) alone, while the opposite side received the same bone graft combined with platelet-rich fibrin (PRF). PRF is a blood-derived material prepared from the patient's own blood and is thought to support tissue healing. The treatment side receiving PRF was determined randomly.

Six months after the sinus lift surgery, dental implants were placed. At that time, small bone samples were collected from the grafted areas. These samples were examined under a microscope to assess new bone formation and the amount of remaining graft material.

The purpose of this study was to determine whether adding PRF to DFDBA improves bone regeneration compared with DFDBA alone during lateral maxillary sinus augmentation.v

DETAILED DESCRIPTION:
This study was designed as a prospective randomized split-mouth clinical investigation to assess bone regeneration following lateral maxillary sinus augmentation using two different grafting approaches.

Patients presenting with bilateral posterior maxillary edentulism and requiring sinus floor elevation prior to dental implant placement were enrolled. Each patient received demineralized freeze-dried bone allograft (DFDBA) alone on one side and DFDBA combined with platelet-rich fibrin (PRF) on the contralateral side, with treatment allocation determined randomly.

All sinus augmentation procedures were performed using a standardized lateral window technique. Platelet-rich fibrin was prepared from autologous venous blood immediately before surgery according to established centrifugation protocols. A fixed healing period of six months was observed prior to implant placement.

During implant surgery, bone core specimens were harvested from the grafted sinus regions using trephine burs. Histologic and histomorphometric analyses were conducted in a blinded manner to quantify tissue composition, including newly formed bone, residual graft material, and connective tissue.

The study aimed to compare the regenerative outcomes of the two grafting strategies and to evaluate the adjunctive role of PRF when combined with an osteoinductive allograft material in lateral maxillary sinus augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years.
* Patients requiring bilateral lateral maxillary sinus augmentation for dental implant placement.
* Adequate residual alveolar bone height allowing for lateral sinus floor elevation.
* Good general health (ASA I or II).
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Presence of systemic diseases affecting bone metabolism (e.g., uncontrolled diabetes, osteoporosis).
* History of head and neck radiotherapy.
* Use of medications known to affect bone healing (e.g., bisphosphonates, corticosteroids).
* Active sinus pathology or chronic sinusitis.
* Heavy smoking (>10 cigarettes per day).
* Pregnancy or lactation.
* Poor oral hygiene or untreated periodontal disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Histomorphometric New Bone Formation (%) | 6 months after lateral maxillary sinus augmentation
  The percentage of newly formed bone in biopsy samples obtained from the augmented maxillary sinus, evaluated by histomorphometric analysis.

SECONDARY OUTCOMES:
Residual Graft Material (%) | 6 months after lateral maxillary sinus augmentation
  The percentage of residual graft material remaining in biopsy samples obtained from the augmented maxillary sinus, assessed by histomorphometric analysis.
Connective Tissue (%) | 6 months after lateral maxillary sinus augmentation
  The percentage of connective tissue present in biopsy samples obtained from the augmented maxillary sinus, evaluated using histomorphometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No